CLINICAL TRIAL: NCT03134742
Title: Prospective Evaluation of Abscopal Radiation Effects on Regional and Distant Bone
Brief Title: Radiation Effects on Bone
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Timothy Damron, M.D., David G. Murray Professor of Orthopedic Surgery, State University of New York - Upstate Medical University
Other Study IDs: 1019460
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Soft Tissue Sarcoma Adult
Keywords: soft tissue sarcoma extremities
MeSH Terms: interventions — Control Groups; Tomography, X-Ray Computed; Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control Group: Subjects will not have any additional scans only those that are standard of care. Their data will be used for comparison
  Interventions: Other: Control Group
- CT Scan only: Three CT Scans will be done of the affected extremity as well as the contralateral extremity at Baseline (pre-radiotherapy), and 6 months and 1 year post-radiotherapy treatment.
  Interventions: Diagnostic Test: CT Scan
- DEXA Scans only: Three DEXA Scans will be done of the affected extremity as well as the contralateral extremity at Baseline (pre-radiotherapy), and 6 months and 1 year post-radiotherapy treatment
  Interventions: Diagnostic Test: DEXA Scans
- CT and DEXA Scans: Three CT Scans and three DEXA Scans will be done of the affected extremity as well as the contralateral extremity at Baseline (pre-radiotherapy), and 6 months and 1 year post-radiotherapy treatment
  Interventions: Diagnostic Test: CT and DEXA Scans

INTERVENTIONS:
Other: Control Group — No interventions this is the control group-no additional scans
  Groups: Control Group
Diagnostic Test: CT Scan — CT Scan of affected and contralateral limb
  Groups: CT Scan only
Diagnostic Test: DEXA Scans — DEXA Scan of affected and contralateral limb
  Groups: DEXA Scans only
Diagnostic Test: CT and DEXA Scans — CT Scan and DEXA Scan of affected and contralateral limb
  Groups: CT and DEXA Scans

SUMMARY:
Post-radiotherapy fragility fractures (caused by weakened bones) are an occasional complication of orthopedic oncology of soft tissue sarcoma patients. Treatment for impending fracture due to radiotherapy does exist in the form of operative stabilization, to prevent the bone from breaking. Without the ability to predict those patients at a higher risk for fracture, indications for treatment are difficult to determine. This study is to determine if there is a correlation between patients undergoing radiotherapy for soft tissue sarcoma and loss of bone density. The study wll evaluate bone loss for short and long term fracture prediction using dual-energy xray, absorptiometry (DEXA [DXA]) and computerized tomography scans (CT Scans)

DETAILED DESCRIPTION:
Post-radiotherapy fragility fractures are a frequent complication of orthopedic oncology care of sarcoma patients, who often receive radiotherapy (XRT) as adjunctive treatment. Prediction of these fractures is difficult as there has been no demonstrable relationship shown, to date, between bone density and fracture risk for this population. Treatment for an impending fracture due to radiotherapy does exist in the form of prophylactic operative stabilization with an intramedullary nail to prevent the bone from breaking. Without the ability to predict those patients at higher risk for fracture, clinical indications for prophylactic treatment are difficult to develop.

Bone density has been investigated as a possible fracture prediction tool. Work by Dhakal et al. suggested specifically that bone density, as measured by dual-energy x-ray absorptiometry (DXA), of the irradiated limb is not decreased following therapeutic doses of radiotherapy (50 Gy) administered for soft tissue sarcomas. However, their technique did not measure pre-radiotherapy bone mineral density (BMD), but rather compared post-radiotherapy BMD of the irradiated site to contralateral and ipsilateral non-irradiated long bones of the extremity. While this technique accounted for disuse osteopenia (bone loss due to decreased use of the afflicted limb), it did not account for any systemic effects of radiation therapy. This is important, because largely based on their work, BMD has not been utilized as a predictor of risk of fracture, and other measures have been sought for this particular clinical situation without success. Others have also failed to show decreased BMD within the irradiated field. However, these studies have either lacked power to show statistical significance or the patient population was pediatric, a growing population in which age related accrual of bone density was a potential confounder.

What Dhakal and others did not account for was the possibility of abscopal (systemic) effects of radiotherapy that might also affect the contralateral and distant sites. Recent work in this investigators laboratory and others using small animal models has suggested that radiation to one limb has statistically significant effects on the contralateral limb in terms of decreased bone mineral density and loss of bone strength. The importance and clinical implications of such an abscopal effect is as of yet unclear. At the very least, its presence calls into question the conclusion that bone density is not decreased at the site of radiation, since differences may only be able to be shown when compared to non-irradiated control subjects. Moreover, there may be an adverse effect on distant bones, further lowering BMD and contributing to fragility fractures, particularly in post-menopausal women who are already at some increased risk. There is mixed clinical data on this topic, with one series of 45,662 prostate cancer patients showing a 76% increased risk of hip fracture (regional bone) following pelvic radiation, but no increased risk of fractures outside the field of radiation in three studies of patients with pelvic radiation for cervical and other female cancers or prostate cancer.

The investigators of this study propose to determine whether human subjects undergoing radiotherapy for soft tissue sarcomas exhibit for abscopal bone loss. Patients in the PI's (Dr. Damron) practice obtain baseline-staging studies, including computerized tomography (CT) of the chest/abdomen/pelvis prior to treatment. Post-treatment, patients then undergo oncology surveillance utilizing routine repetitive computerized tomography of the chest and sometimes of the abdomen/pelvis for a subset where the baseline abdomen/pelvis CT scans show abnormalities that need to be followed. These CT scans, when combined with calibration phantoms of known density, afford a prime opportunity to quantify bone mineral density based on those scans at sites distant to the primary site of radiotherapy (typically in the extremity).

This project will also evaluate a secondary aim, that of comparing effectiveness of utilization of CT vs BMD as a tool to evaluate bone loss in short term with a potential for long term fracture prediction in this patient population. In order to accomplish this aim, simultaneously, in a subset of patients who give consent for non-standard of care DXA scans, the investigators will evaluate the potential abscopal bone loss by assessing changes in BMD as measured by DXA, a tool that is a gold standard for bone density evaluation and for fracture prediction in routine clinical practice. The investigators will compare BMD pre- and post-radiotherapy at the site of irradiation, and further compare this change to that of the change in BMD at distant sites.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Dr. Damron's being treated for soft tissue sarcoma of an extremity, who will undergone radiotherapy, and will follow with Dr. Damron for routine oncology surveillance with routine CT scans of the chest at minimum.
* Must be at least 18 years of age and no older than 89 years of age.

Exclusion Criteria:

* Patients who are treated with radiotherapy but who do not have soft tissue sarcoma, such as those with metastatic carcinoma,
* Patients who have soft tissue sarcoma who will not receive adjuvant radiotherapy, such as those with atypical lipomatous tumors or other low grade soft tissue sarcomas
* Patients who will not be obtaining their follow up CT studies at Upstate Bone and Joint Center-since the calibration phantom needs to be located in one central location.
* Incarcerated patients
* Patients younger than 18 years of age

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects between the ages of 18 and 89 years of age, who have been diagnosed with soft tissue sarcoma of an extremity, who have not had radiotherapy treatment, or been diagnosed with metastatic carcinoma, atypical lipomatous tumors or low grade soft tissue sarcomas.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-03-13 (Actual); Primary Completion 2025-04-13 (Estimated); Study Completion 2025-04-13 (Estimated)

PRIMARY OUTCOMES:
Determine whether subjects undergoing radiotherapy for soft tissue sarcoma exhibit abscopal bone loss | 12 months post radiation
  CT Scans combined with calibration phantoms will be used to quantify bone density, when compare pre- and post-radiotherapy at the site of irradiation and at distant sites (contralateral limb)

SECONDARY OUTCOMES:
Comparing effectiveness of utilization of CT vs DEXA as a tool to evaluate bone loss in short term with potential for long term fracture prediction | 12 months post radiation
  DEXA Scans will be used to evaluate the potential abscopal bone loss by assessing changes in bone mineral density as measured by DEXA, when compared pre- and post-radiotherapy at the site of irradiation and at distant sites (contralateral limb)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Damron, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No